CLINICAL TRIAL: NCT03888027
Title: A Randomized Controlled Trial of a Volunteer-driven Walking Intervention to Improve Hospital-associated Deconditioning and Frailty
Brief Title: WalkMORE: A Volunteer-driven Walking Intervention
Acronym: WalkMORE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 prevented volunteers from entering and interacting with patients. The study intervention was reliant on volunteers engagin directly with participants.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ReDA 6072
Record Dates: First submitted 2019-03-13; First posted 2019-03-25 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-03

CONDITIONS: Frailty; Deconditioning; Early Ambulation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Patients will be randomized via REDCap (Research Electronic Data Capture), a secure, centralized web-based randomization module to:
  1. Standard of care; or
  2. WalkMORE Ambulation program + Standard of care. Patients will ambulate with a trained WalkMORE Volunteer Coach two times per day; once in the morning (0900-1200hrs) and once in the afternoon (1300-1700hrs), Monday- Friday, until hospital discharge. Patients randomized to the WalkMORE intervention will be assessed daily by the Research Coordinator to ensure patients remain fit for independent ambulation. The duration of each walking session will be determined daily by the RC and the medical team.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients receive no intervention
- WalkMORE group (Active Comparator): Patients will be randomized via REDCap (Research Electronic Data Capture), a secure, centralized web-based randomization module to:
  1. Standard of care; or
  2. WalkMORE Ambulation program + Standard of care. Patients will ambulate with a trained WalkMORE volunteer two times per day; once in the morning (0900-1200hrs) and once in the afternoon (1300-1700hrs), Monday- Friday, until hospital discharge. Patients randomized to the WalkMORE intervention will be assessed daily by the Research Coordinator to ensure patients remain fit for independent ambulation. The duration of each walking session will be determined daily by the RC and the medical team.
  Interventions: Behavioral: WalkMORE group

INTERVENTIONS:
Behavioral: WalkMORE group — Hospitalized Internal Medicine patients will walk with trained volunteers twice daily until hospital discharge.
  Arms: WalkMORE group

SUMMARY:
Patients admitted to hospital typically experience periods of decreased activity or bed-rest. This reduced activity level leads to deconditioning - a loss of muscle mass, muscle strength (by 2-5% per day), and muscle shortening. Even among patients who were ambulatory at the time of admission, deconditioning has been linked with deleterious effects, such as increased rates of falls, functional decline, and frailty. Furthermore, it has been suggested that the physiological stresses associated with hospitalization - including deconditioning, as well as sleep deprivation and poor nutrition - makes discharged patients vulnerable to recurrent or new illnesses and to frailty. This physiological stress-induced vulnerability has been coined "post-hospital syndrome" and is thought to have a role in most hospital readmissions. The investigators hypothesize that by engaging ambulatory patients to walk with trained volunteers, patients will increase their amount of walking, have less deconditioning and functional decline, and consequently, fewer falls. Furthermore, the investigators anticipate that patients who walk with a trained volunteer will have reduced length-of-stay in hospital and decreased likelihood of readmission. Finally, as shown in other similar programs, the investigators anticipate an overall improvement in the patient experience. The investigator's novel initiative focuses on a single, volunteer-based intentional ambulation program that can deliver the benefits of early mobility in a cost-effective way. The program design engages trained volunteers to increase patient ambulation in a way that both increases patient mobility and reduces healthcare professionals' workload.

DETAILED DESCRIPTION:
WalkMORE is a single-center randomized controlled trial. The investigators will enroll up to 800 ambulatory patients admitted to the Internal Medicine unit (located on the 4th floor of University Hospital) who are >18 years of age and are anticipated to require a >48 hour hospital admission. A maximum of 6 patients will be assigned to each treatment arm at any given time. The investigators will recruit patients into the WalkMORE program over a 2 year period. The research coordinator (RC) will screen patients admitted to the Internal Medicine unit in the preceding 24-hour period to identify patients who fulfill the eligibility criteria. Patients will be randomized via REDCap (Research Electronic Data Capture), a secure, centralized web-based randomization module to:

1. Standard of care; or
2. WalkMORE Ambulation program + Standard of care. Patients will ambulate with a trained WalkMORE Volunteer two times per day; once in the morning (0900-1200 hrs) and once in the afternoon (1300-1600 hrs), Monday- Friday, until hospital discharge. Patients randomized to the WalkMORE intervention will be assessed daily by the RC to ensure patients remain fit for independent ambulation. The duration of each walking session will be determined daily by the RC and the medical team.

After obtaining written informed consent from eligible patients the RC will randomize patients, collect demographics and hospital admission details from patients' hospital charts and perform the Barthel Index and complete the Charlson Comorbidity Index (CCI) for all patients. The Barthel Index (BI) measures the extent to which patients can function independently and has mobility in their activities of daily living (ADL). The Charlson Comorbidity Index categorizes and scores the comorbidities of patients. The CCI can be used to predict short term and long-term outcomes such as function, hospital length of stay and mortality rates. The CCI will be completed using information gathered from patients' hospital chart.with all patients.

All patients will be assigned a scientific pedometer on the day of randomization. The modus Health StepWatch™ is an activity monitor worn on the ankle via a velcro strap. It is a small, lightweight device that will count and record patients' steps throughout hospital stay, ending at hospital discharge. Research personnel will be responsible for fitting the StepWatch monitor to patients' ankle. The device is smaller than a deck of cards (7.5 x 5.0 x 2.0 cm) and weighs 38 grams.

Frailty and de-conditioning will be measured on Study Day 3. Frailty will be assessed using the Jamar Hand Dynamometer. Patients are instructed to squeeze the handle of the instrument with their maximum force for three seconds; the peak-hold (in kilograms) is recorded on the instrument. Three successive peak-hold measurements will be recorded. The device measures 10 x 20 x 33cm and weighs 1.3 kg. Deconditioning will be measured using the Timed Up and Go (TUG) test, patients will be asked to stand up from a chair, walk three metres, turn around, and walk back to the chair and sit.

After hospital discharge the RC will follow up with patients for 2 brief telephone interviews. On the third day after discharge, Patient Satisfaction surveys will be conducted by the RC to assess patient satisfaction with their hospital experience and with the WalkMORE program. On day 30 after randomization, the RC will contact patients to conduct a brief interview consisting of: a health status survey (EQ-5D), a functional status assessment (Barthel Index) and to collect data regarding clinical outcomes (ER visits, re-hospitalizations, and falls). Each telephone interview is expected to last approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and appropriate for independent ambulation (with or without gait aids) as determined daily by the health care team
2. Cognitively safe for participation
3. Anticipated to remain hospitalized ≥48 hours
4. Inpatient, admitted to Internal Medicine at University Hospital
5. Age >18 years

Exclusion Criteria:

1. Preexisting condition precludes patient from independent ambulation at time of admission
2. Active medical condition precludes patient from safely participating
3. Preexisting condition or active medical condition renders patient unfit to participate as judged by the admitting team
4. Patients who refuse to participate or are unable to provide informed consent.
5. Communication barrier (due to hearing/vision impairment, or language barrier)
6. Patients receiving treatment from an LHSC inpatient Physiotherapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Re-hospitalization | 30 days after randomization
  Number of patients re-admitted to hospital
Presentation to emergency department | 30 days after randomization
  Number of patients seen in the hospital emergency department
Prolonged index hospital admission | 30 days after randomization
  Number of patients with extended length of hospital admission

SECONDARY OUTCOMES:
Length of stay for index hospital admission | 30 days after randomization
  Number of days patient was hospitalized
Post-discharge Falls | 30 days after randomization
  Composite of number of readmissions and emergency room visits secondary to patients experiencing a fall post-discharge
Timed-Up-And-Go | 30 days after randomization
  Measure of de-conditioning between the two study arms using
Barthel Index | 30 days after randomization
  ordinal scale used to measure performance in activities of daily living. Minimum score is zero and maximum score is 100, higher score represent better outcomes.
Frailty | 30 days after randomization
  Measure of frailty between the two study arms using the Jamar Hand Dynamometer data
Deconditioning | 30 days after randomization
  total steps as measured by pedometer as a measure of deconditioning
Increased number of steps | 30 days after randomization
  proportion of patients who increase step count by 200 steps per day
EQ-5D | 30 days after randomization
  A STANDARDIZED INSTRUMENT FOR USE AS A MEASURE OF HEALTH OUTCOME. The EQ-VAS scale ranges from a minimum of zero and a maximum of 100 and is the participants subjective score of how good or poor their health is at the time the scale is presented to them. Higher values represent a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- LHSC-University Hospital, London, Ontario, Canada